CLINICAL TRIAL: NCT01505608
Title: A Randomized, Phase I/II Trial of Irinotecan and Temozolomide Compared to Irinotecan and Temozolomide in Combination With TPI 287 in Patients With Primary Refractory or Early Relapsed Neuroblastoma
Brief Title: Randomized Efficacy Study of TPI 287 to Treat Primary Refractory or Early Relapsed Neuroblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Giselle Sholler (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Vice Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC 005
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — TPI-287; Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A- Temozolomide and Irinotecan (Active Comparator): 1. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  2. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  Patients who show progression on the I+TMZ arm may crossover to the I+TMZ+TPI 287 arm at anytime during cycles 1 to 6. If there is evidence of progression after completion of the I+TMZ arm (after completion of cycle 6) then the patient will have been considered to have completed therapy and is not eligible for the crossover.
  Interventions: Drug: Temozolomide; Drug: Irinotecan
- Arm B- Temozolomide/Irinotecan + TPI 287 (Experimental): Cycle 1 to 6: Irinotecan and Temozolomide in combination with TPI 287
  1. Intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  2. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  3. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  Interventions: Drug: TPI 287; Drug: Temozolomide; Drug: Irinotecan

INTERVENTIONS:
Drug: TPI 287 — Subjects will receive six cycles of intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  Arms: Arm B- Temozolomide/Irinotecan + TPI 287
Drug: Temozolomide — Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle
  Other Names: temodar
Drug: Irinotecan — Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.

SUMMARY:
The purpose of this research study is to evaluate a new investigational drug (TPI 287) for early relapsed neuroblastoma. An investigational drug is one that has not yet been approved by the Food and Drug Administration. This investigational drug is called TPI 287. This study will look at the tumor's response to the study drug, TPI 287, in combination with Irinotecan and Temozolomide versus the combination of Irinotecan and Temozolomide alone. This study will also evaluate the safety and tolerability of the study drug, TPI 287.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically proven Neuroblastoma and confirmation of primary refractory or recurrent disease with histologic confirmation at diagnosis or at the time of recurrence/progression. Subjects must have primary refractory or have early relapse disease (early relapse disease is defined as having received ≤ one or two relapse therapies).
* Subjects must be age >12 months and diagnosed before the age of 21 years
* Measurable disease, including at least one of the following:

Measurable tumor >10 mm by CT or MRI Positive bone marrow biopsy/aspirate Positive MIBG

* Current disease state must be one for which there is currently no known curative therapy
* Lansky Play Score or Karnofsky scale must be more than 30
* Subjects without bone marrow metastases must have an ANC > 750/μl and platelet count >50,000/μl
* Adequate Renal Function Defined As Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 or
* A serum creatinine based on age/gender table
* Adequate liver function must be demonstrated, defined as:

Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age SGPT (ALT) < 10 x upper limit of normal (ULN) for age SGOT (AST) < 10x upper limit of normal (ULN) for age

* No other significant organ toxicity defined as >Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE V4.0- http://ctep.cancer.gov/forms/CTCAEv4.pdf)
* A negative urine pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Informed Consent: All subjects and/or legal guardians must sign written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines
* Subjects may have received microtubulin inhibitors during previous therapies.
* Subjects may have received any number of prior biological therapies.

Exclusion Criteria:

* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the effects of prior chemotherapy (hematological and bone marrow suppression effects), generally at least 3 weeks from the most recent administration (6 weeks for nitrosoureas). Subjects may not have received more than 1 cycle of Irinotecan and Temozolomide as previous relapse therapy.
* Subjects who have received any myeloablative therapy within the previous 2 months.
* Subjects receiving any investigational drug concurrently
* Subjects with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 (NCI CTCAE V4.0), or active, serious infections requiring parenteral antibiotic therapy.
* Subjects with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a subject's ability to sign or the legal guardian's ability to sign the informed consent, and subject's ability to cooperate and participate in the study
* Subjects with known hypersensitivity to any of the components of the drugs to be administered on study.
* Subjects who have previously been treated with TPI 287.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Eslin, MD, Study Chair — Arnold Palmer Hospital for Children
Locations (8):
- United States (8):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children- MD Anderson, Orlando, Florida
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina

REFERENCES:
- See also: Beat Childhood Cancer — https://beatcc.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1- All patients assigned to TPI 287 group. Randomization began in Phase 2- Arm A patients were allowed to cross over to Arm B during cycles 1-6 if they experienced progression. 0 (zero) Arm A patients crossed over to Arm B on this study.
Groups:
- Arm A- Temozolomide and Irinotecan: 1. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  2. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  During Phase 2- Patients who show progression on the I+TMZ arm may crossover to the I+TMZ+TPI 287 arm at anytime during cycles 1 to 6. If there is evidence of progression after completion of the I+TMZ arm (after completion of cycle 6) then the patient will have been considered to have completed therapy and is not eligible for the crossover.
  Temozolomide: Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle
  Irinotecan: Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
- Arm B- Temozolomide/Irinotecan + TPI 287: Cycle 1 to 6: Irinotecan and Temozolomide in combination with TPI 287
  1. Intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  2. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  3. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  TPI 287: Subjects will receive six cycles of intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  Temozolomide: Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle
  Irinotecan: Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
Period: Phase I
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287
Started | 0 (Randomization to Arm A began in Phase 2. All patients in Phase I were enrolled to receive TPI 287.) | 8
Completed | 0 | 2
Not Completed | 0 | 6
Not completed — Lack of Efficacy | 0 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Phase II
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287
Started | 2 (Phase 2 was new enrollment, not the same patients from Phase 1.) | 4 (Phase 2 was new enrollment, not the same patients from Phase 1.)
Completed | 0 | 2
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A- Temozolomide and Irinotecan: 1. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  2. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  Patients who show progression on the I+TMZ arm may crossover to the I+TMZ+TPI 287 arm at anytime during cycles 1 to 6. If there is evidence of progression after completion of the I+TMZ arm (after completion of cycle 6) then the patient will have been considered to have completed therapy and is not eligible for the crossover.
  Temozolomide: Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle
  Irinotecan: Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287 | Total
Number analyzed (Participants) | 2 | 12 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 11 | 13
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 9 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 12 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 2 | 8 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To determine the safety and tolerability of TPI 287 in combination with Irinotecan and Temozolomide (TPI+I+TMZ) in pediatric and young adult patients with primary refractory or recurrent Neuroblastoma.
  Phase I patients were all enrolled to receive TPI 287. Phase 2 is where randomization began. Patients were different patients than the Phase 1 patients. Below all patients that received TPI 287 are included in the TPI 287 group. This includes Phase I patients and the Phase 2 patients randomized to TPI 287.
Time Frame: 6 months
Population: This group includes the 8 patients enrolled to phase 1 TPI 287 portion of the study plus the 4 additional patients randomized to TPI 287 in the Phase 2 portion = 12 patients total that received TPI 287 on this study.
Measure: Number; unit: participants
Groups:
- TPI 287: Cycle 1 to 6: Irinotecan and Temozolomide in combination with TPI 287
  1. Intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  2. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  3. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  TPI 287: Subjects will receive six cycles of intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  Temozolomide: Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle
  Irinotecan: Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
- Arm A- TMZ + Irinotecan Only: Did not receive TPI 287
Arm/Group | TPI 287 | Arm A- TMZ + Irinotecan Only
Number analyzed (Participants) | 12 | 2
participants | 7 | 0

2. Primary Outcome: Overall Response Rate (ORR) of Participants Using RECIST Criteria
Description: Phase I portion of trial- All patients enrolled to recieve TPI+I+TMZ. These patients will be added to the Phase II patients that were randomized to Arm B- Arm with TPI 287 (recieved same tx as Phase I participatns).
  Phase II portion of trial- TPatients enrolled to this portion (different patients than enrolled to Phase 1) were randomized to Arm A: I+TMZ OR Arm B: TPI+I+TMZ Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 3 years
Population: 8 enrolled to Phase 1: two were non-evaluable =6 move to analysis. Another 4 randomized to Arm B with TPI 287 in Phase 2=10 evaluable in TPI 287 analysis.
  2 subjects were enrolled in the Phase 2 randomized portion of the trial to Arm A- without TPI 287. This makes 2 evaluable subjects in this analysis population (did not receive TPI 287).
Measure: Number; unit: participants
Groups:
- Phase I Patients + Phase II Assigned Arm B- Tmz +I+ TPI 287: Cycle 1 to 6: Irinotecan and Temozolomide in combination with TPI 287
  1. Intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  2. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  3. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
  TPI 287: Subjects will receive six cycles of intravenous (IV) TPI 287 at a dose of 125 mg/m2 on Days 1, 8 and 15 of a 28-day cycle.
  Temozolomide: Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle
  Irinotecan: Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
Arm/Group | Arm A- Temozolomide and Irinotecan | Phase I Patients + Phase II Assigned Arm B- Tmz +I+ TPI 287
Number analyzed (Participants) | 2 | 10
participants | 0 | 2

3. Secondary Outcome: Pharmacokinetics (PK) of TPI 287 in the Phase I Population of This Trial.
Description: To evaluate the drug levels and pharmacokinetics (PK) of TPI 287 from blood samples at multiple time points within the first 24 hours on study.
Time Frame: 1 year
Population: PK's not run due to early closure of study. Data not collected or analyzed threfore no data exists.
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measure Quality of Life of Children Receiving TPI287 Using PedsQL Questionnaires
Description: Evaluate the impact on QOL of children receiving TPI+I+TMZ
Time Frame: 3 years
Population: QOL's not collected due to early closure of study. Data not collected or analyzed threfore no data exists.
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS) of Participants Using Days Until Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years
Population: Arm A- 2 subjects randomized to TMZ+I. Arm B- 6 evalubale patients in Phase 1 + 4 evaluable patients in Phase 2- all received TMZ+I+TPI
Measure: Number; unit: Days
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287
Number analyzed (Participants) | 2 | 10
Days | 22 | 125

6. Secondary Outcome: Median Overall Survival (OS) of Participants
Description: To determine OS and clinical benefit (CR/PR/SD) in this population
Time Frame: 3 years
Population: Not evaluated due to early closure. Study data does not exist.
Arm/Group | Arm A- Temozolomide and Irinotecan | Arm B- Temozolomide/Irinotecan + TPI 287
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: New adverse events collected from first dose of study drug to 30 days past last dose of study drug. Related adverse events followed until resolution, approximately 1 year.
Groups:
- Phase II Arm A- Subjects That Did Not Receive TPI 287: Cycle 1 to 6: Irinotecan and Temozolomide
  1. Oral (PO) Temozolomide at a dose of 100mg/m2 on days 1-5 of each 28 day cycle.
  2. Intravenous (IV) Irinotecan at a dose of 10mg/m2 on days 1-5 and 8-12 of each 28 day cycle.
Arm/Group | TPI 287 | Phase II Arm A- Subjects That Did Not Receive TPI 287
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/2
Other Adverse Events (participants affected / at risk) | 11/12 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 (N=12) | Phase II Arm A- Subjects That Did Not Receive TPI 287 (N=2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Progression of Disease resulting in Death (General disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TPI 287 (N=12) | Phase II Arm A- Subjects That Did Not Receive TPI 287 (N=2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Infusion Related Reaction (General disorders) | 4 (16) | 0 (0)
lymphocytopenia (Blood and lymphatic system disorders) | 2 (21) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (18) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 3 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less